CLINICAL TRIAL: NCT02643082
Title: A Randomized, Double-Blind, Two Treatment, Two Period, Chronic Dosing (2 Weeks), Cross-Over, Single-Center Study to Evaluate the Effects of PT003 and Placebo MDI on Specific Image Based Airway Volumes and Resistance in Subjects With Moderate to Severe COPD
Brief Title: A Study to Assess the Effects of PT003 and Placebo MDI on Specific Image Based Airway Volumes and Resistance in Subjects With Moderate to Severe COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PT003018; NCT03024346 (obsolete NCT alias)
Record Dates: First submitted 2015-12-10; First posted 2015-12-30 (Estimated); Results first posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-02

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- GFF MDI, 14.4/9.6μg (Experimental): Glycopyrronium and Formoterol Fumarate Inhalation Aerosol; PT003, Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler (GFF MDI)
  Interventions: Drug: GFF MDI (PT003) 14.4/9.6μg
- Placebo MDI (Placebo Comparator): Placebo Metered Dose Inhaler (MDI)
  Interventions: Drug: Placebo MDI

INTERVENTIONS:
Drug: GFF MDI (PT003) 14.4/9.6μg — Glycopyrronium and Formoterol Fumarate
  Other Names: GFF
  Arms: GFF MDI, 14.4/9.6μg
Drug: Placebo MDI — Comparator: Placebo MDI which contains no active ingredients
  Other Names: Placebo
  Arms: Placebo MDI

SUMMARY:
Study to Evaluate the Effects of PT003 and Placebo MDI on Specific Image Based Airway Volumes and Resistance With Moderate to Severe COPD.

DETAILED DESCRIPTION:
Enrolled patients with COPD who were randomized to receive either PT003 MDI or Placebo MDI first and then crossed over to receive the opposite intervention. The study consisted of 2 treatment periods of 14 days separated by a washout period of 5-21 days.

ELIGIBILITY:
Inclusion Criteria:

* Non-child bearing potential (ie, physiologically incapable of becoming pregnant, including any female who is 2 years post-menopausal); or Child bearing potential, has a negative urine pregnancy test at Visit 1 and agrees to an acceptable method of contraception
* Subjects with an established clinical history of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS)
* Current or former smokers with a history of at least 10 pack-years of cigarette smoking.
* At Visit 1, FEV1/FVC ratio must be <0.70
* At Visit 1, post-bronchodilator FEV1/FVC ratio of <70% and FEV1 must be 30% to 80% before predicted normal value, calculated using NHANES III reference equations.

Exclusion criteria:

* Significant diseases other than COPD, i.e., disease or condition which, in the opinion of the Investigator, may put the subject at risk because of participation in the study or may influence either the results of the study or the subject's ability to participate in the study.
* Women who are pregnant or lactating, or are planning to become pregnant during the course of the study, or women of childbearing potential who are not using an acceptable method of contraception.
* Subjects, who in the opinion of the Investigator, have a current diagnosis of asthma.
* Subjects who have been hospitalized due to poorly controlled COPD within 3 months prior to Visit 1 (Screening) or during the run-in period (Visit 1 to Visit 2).
* Subjects who have poorly controlled COPD, defined as acute worsening of COPD that requires treatment with oral corticosteroids or antibiotics within 6 weeks prior to Visit 1 (Screening) or during the run-in period (Visit 1 to Visit 2).
* Subjects with a diagnosis of angle closure glaucoma will be excluded, regardless of whether or not they have been treated.
* Subjects who have a history of hypersensitivity to β2-agonists, glycopyrronium or other muscarinic anticholinergics, or any component of the MDI.

Please refer to the study protocol for the complete inclusion criteria list.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2017-01-26 (Actual); Study Completion 2017-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chad Orevillo, Study Director — Pearl Therapeutics
Locations (1):
- Research Site, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
AstraZeneca's policy is to share data with researchers if the request is in scope of our policy. The policy and additional information can be found on astrazenecaclinicaltrials.com.

REFERENCES:
- [Derived] De Backer W, De Backer J, Vos W, Verlinden I, Van Holsbeke C, Clukers J, Hajian B, Siddiqui S, Jenkins M, Reisner C, Martin UJ. A randomized study using functional respiratory imaging to characterize bronchodilator effects of glycopyrrolate/formoterol fumarate delivered by a metered dose inhaler using co-suspension delivery technology in patients with COPD. Int J Chron Obstruct Pulmon Dis. 2018 Aug 30;13:2673-2684. doi: 10.2147/COPD.S171707. eCollection 2018. PMID 30214185
- See also: Protocol with updated PDFA coverpage — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4142&filename=PT003018-Protocol-Redacted%20updated%20with%20coverpage%20PDFA.pdf
- See also: Updated version per comments from CT.gov — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4142&filename=PT003018-Protocol-Redacted%20updated%20with%20coverpage%20PDFA.pdf
- See also: Updated version per CT.gov comments — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4142&filename=PT003018-12-1-09-statistical-methods-and-analysis-sap_Redacted%2020180524.pdf
- See also: Updated version per CT.gov comments — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4142&filename=PT003018%20updated%20statistical-methods-and-analysis-sap_Redacted%2020180924.pdf
- See also: Updated version per comments from CT.gov — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4142&filename=PT003018%20Protocol%20Cover%20page%20updated%2020180924.pdf
- See also: Updated version per CT.gov comments — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4142&filename=PT003018-12-1-09-statistical-methods-and-analysis-sap-Redacted-PDFA.pdf
- See also: Updated version per comments from CT.gov — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4142&filename=PT003018-Protocol-Redacted-PDFA.pdf
- See also: Updated version per comments from CT.gov — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4142&filename=PT003018-02MAY2016-Protocol-Redacted-PDFA.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 1 site in Antwerp Belgium from January 2016 to December 2016.The study was anticipated to run for approximately 9 months but not to expected to exceed 12 months. The study period was duration was expected to run approximately 13 weeks for each subject.
Pre-assignment Details: Subjects were randomized into 1 of 2 treatment sequences: subjects in Sequence 1 received GFF MDI in Treatment Period 1 followed by Placebo MDI in Treatment Period 2, and subjects in Sequence 2 received Placebo MDI in Treatment Period 1 followed by GFF MDI in Treatment Period 2. There was a a washout of 5-21 days,in between treatment periods.
Groups:
- GFF MDI/Placebo MDI: Treatment Sequence of Glycopyrronium Formoterol Fumarate Metered Dose Inhalation/Placebo Metered Dose Inhalation
- Placebo MDI/GFF MDI: Treatment Sequence of Placebo Metered Dose Inhalation/Glycopyrronium Formoterol Fumarate Metered Dose Inhalation
Period: Period 1
Arm/Group | GFF MDI/Placebo MDI | Placebo MDI/GFF MDI
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Washout
Arm/Group | GFF MDI/Placebo MDI | Placebo MDI/GFF MDI
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0
Period: Period 2
Arm/Group | GFF MDI/Placebo MDI | Placebo MDI/GFF MDI
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: ITT Population - all subjects who were randomized to treatment. Treatment was assigned as randomized regardless of the treatment actually received.
Groups:
- Overall Study: All Randomized Patients
Arm/Group | Overall Study
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.8 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Specific Airway Volume (siVaw)
Description: Specific image-based airway volume. Average across lobe, adjusted for lobe volume
Time Frame: Day 15
Population: ITT Population
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mL/L
Groups:
- GFF MDI 14.4/9.6 µg: GFF MDI
- Placebo MDI: Placebo
Arm/Group | GFF MDI 14.4/9.6 µg | Placebo MDI
Number analyzed (Participants) | 20 | 19
mL/L | 1.79 [1.48 to 2.16] | 1.02 [0.85 to 1.24]
Statistical Analysis 1: Comparison: GFF MDI 14.4/9.6 µg vs Placebo MDI; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean ratio between treatments = 1.75, 95% CI 2-sided [1.65 to 1.86]

2. Secondary Outcome: Airway Resistance (iRaw)
Description: iRaw represents the airway resistance, averaged across lobes, without correction for lung lobe volume
Time Frame: Day 15
Population: ITT Population
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: kPa s/L
Arm/Group | GFF MDI 14.4/9.6 µg | Placebo MDI
Number analyzed (Participants) | 20 | 19
kPa s/L | 0.07 [0.06 to 0.10] | 0.25 [0.19 to 0.33]
Statistical Analysis 1: Comparison: GFF MDI 14.4/9.6 µg vs Placebo MDI; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean ratio between treatments = 0.29, 95% CI 2-sided [0.26 to 0.33]

3. Primary Outcome: Specific Airway Resistance (siRaw)
Description: Specific image-based airway resistance. Average across lobes, adjusted for lobe volume
Time Frame: Day 15
Population: ITT Population
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: kPa s
Arm/Group | GFF MDI 14.4/9.6 µg | Placebo MDI
Number analyzed (Participants) | 20 | 19
kPa s | 0.09 [0.07 to 0.11] | 0.30 [0.23 to 0.40]
Statistical Analysis 1: Comparison: GFF MDI 14.4/9.6 µg vs Placebo MDI; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean ratio between treatments = 0.29, 95% CI 2-sided [0.25 to 0.33]

4. Secondary Outcome: Airway Volume (iVaw)
Description: iVaw represents the airway Volume, averaged across lobes, without correction for lung lobe volume
Time Frame: Day 15
Population: ITT Population
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | GFF MDI 14.4/9.6 µg | Placebo MDI
Number analyzed (Participants) | 20 | 19
mL | 2.11 [1.73 to 2.58] | 1.18 [0.97 to 1.44]
Statistical Analysis 1: Comparison: GFF MDI 14.4/9.6 µg vs Placebo MDI; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean ratio between treatments = 1.79, 95% CI 2-sided [1.67 to 1.92]

5. Secondary Outcome: Change From Baseline in FEV1 (L) at Day 15
Description: Change from baseline in Forced Expiratory Volume at 1 second
Time Frame: Baseline and Day 15
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI 14.4/9.6 µg | Placebo MDI
Number analyzed (Participants) | 20 | 19
Liters | 0.334 [0.245 to 0.422] | -0.110 [-0.198 to -0.022]
Statistical Analysis 1: Comparison: GFF MDI 14.4/9.6 µg vs Placebo MDI; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean Difference Between Treatments = 0.443, 95% CI 2-sided [0.318 to 0.569]

6. Secondary Outcome: Change From Baseline in FRC (L) at Day 15
Description: Change from baseline in Functional Residual Capacity
Time Frame: Baseline and Day 15
Population: ITT Population
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI 14.4/9.6 µg | Placebo MDI
Number analyzed (Participants) | 20 | 19
Liters | 0.90 [0.86 to 0.93] | 1.03 [0.99 to 1.07]
Statistical Analysis 1: Comparison: GFF MDI 14.4/9.6 µg vs Placebo MDI; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean ratio between treatments = 0.87, 95% CI 2-sided [0.82 to 0.92]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject signed consent throughout the two treatment periods and washout period (approximately 49 days) and up to 10 days following the last dose of study drug.
Description: The Safety Population was defined as all subjects who were randomized to treatment regardless and received at least one dose of study treatment. Serious adverse events collected from the time the subject signed consent up to 14 days following the last dose of study drug.
Arm/Group | Overall Study | GFF MDI 14.4/9.6 µg | Placebo MDI
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 2/20 | 1/20 | 1/19
Other Adverse Events (participants affected / at risk) | 15/20 | 12/20 | 8/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=20) | GFF MDI 14.4/9.6 µg (N=20) | Placebo MDI (N=19)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=20) | GFF MDI 14.4/9.6 µg (N=20) | Placebo MDI (N=19)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Obstructive Airway Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 2 (2) | 1 (1)
Tremor (Nervous system disorders) | 2 (3) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 1 (1) | 0 (0)
Iron Defficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Renal Mass (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal Pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent it's opinions, or the opinions of the publication committee, if these differ with the proposed publication.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-02-27): https://cdn.clinicaltrials.gov/large-docs/82/NCT02643082/SAP_000.pdf
  • Study Protocol (2016-05-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT02643082/Prot_001.pdf